CLINICAL TRIAL: NCT00660179
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group, Event-driven, Phase III Study to Assess the Effects of Macitentan (ACT-064992) on Morbidity and Mortality in Patients With Symptomatic Pulmonary Arterial Hypertension
Brief Title: Study of Macitentan (ACT-064992) on Morbidity and Mortality in Patients With Symptomatic Pulmonary Arterial Hypertension
Acronym: SERAPHIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-055-302
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension SERAPHIN
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Macitentan (ACT-064992) tablet, 3 mg, once daily
  Interventions: Drug: macitentan (ACT-064992)
- 2 (Experimental): Macitentan (ACT-064992) tablet, 10 mg, once daily
  Interventions: Drug: macitentan (ACT-064992)
- 3 (Placebo Comparator): Matching placebo, once daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: macitentan (ACT-064992) — Tablet, 3 mg dosage, once daily
  Arms: 1
Drug: macitentan (ACT-064992) — Tablet, 10 mg dosage, once daily
  Arms: 2
Drug: placebo — Matching placebo, once daily
  Arms: 3

SUMMARY:
The AC-055-302/SERAPHIN study will be an event-driven Phase III study, comparing two different doses of macitentan (ACT-064992) (3 and 10 mg) vs placebo in patients with symptomatic PAH. The main study objective is to demonstrate that macitentan (ACT-064992) prolongs time to the first morbidity or mortality event, and to evaluate the benefit/risk profile of macitentan (ACT-064992) in the treatment of patients with symptomatic PAH.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study mandated procedure.
2. Patients with symptomatic pulmonary arterial hypertension (PAH) in modified World Health Organization (WHO) functional class II to IV.
3. Patients with the following types of pulmonary arterial hypertension (PAH) belonging to groups 1.1 to 1.3 of the Venice classification:

   * Idiopathic (IPAH);
   * Familial (FPAH); or
   * Related to:

     * Collagen vascular disease;
     * Simple, congenital systemic-to-pulmonary shunts at least 1 year post surgical repair;
     * Human immunodeficiency virus (HIV) infection; or
     * Drugs and toxins.
4. PAH diagnosis confirmed by hemodynamic evaluation performed prior to randomization and showing all of the following:

   * Mean pulmonary artery pressure (mPAP) > 25 mmHg at rest;
   * Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) < 15 mmHg; and
   * Pulmonary vascular resistance (PVR) at rest >= 320 dyn×sec/cm^5.
5. 6-minute walk distance (6MWD) >= 50 m.
6. Men or women > 12 years of age (women of childbearing potential must have a negative pre-treatment serum pregnancy test and must use a reliable method of contraception).

Exclusion Criteria:

1. PAH associated with portal hypertension, thyroid disorders, glycogen storage disease, Gaucher''s disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders or splenectomy.
2. PAH associated with non corrected simple congenital systemic-to-pulmonary shunts, and combined and complex systemic-to-pulmonary shunts, corrected or non corrected.
3. PAH associated with significant venous or capillary involvement (PCWP > 15 mmHg), known pulmonary veno-occlusive disease, and pulmonary capillary hemangiomatosis.
4. Persistent pulmonary hypertension of the newborn.
5. Pulmonary Hypertension belonging to groups 2 to 5 of the Venice classification.
6. Moderate to severe obstructive lung disease: forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) < 70% and FEV1 < 65% of predicted value after bronchodilator administration.
7. Moderate to severe restrictive lung disease: total lung capacity (TLC) < 60% of predicted value.
8. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C.
9. Estimated creatinine clearance < 30 mL/min
10. Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.5 times the upper limit of normal.
11. Hemoglobin < 75% of the lower limit of the normal range.
12. Systolic blood pressure < 100 mmHg.
13. Acute or chronic physical impairment (other than dyspnea), limiting the ability to comply with study requirements.
14. Pregnant or breast-feeding.
15. Known concomitant life-threatening disease with a life expectancy < 12 months.
16. Body weight < 40 kg.
17. Any condition that prevents compliance with the protocol or adherence to therapy.
18. Recently started (< 8 weeks prior to randomization) or planned cardio-pulmonary rehabilitation program based on exercise.
19. Treatment with endothelin receptor antagonists (ERAs) within 3 months prior to randomization.
20. Systemic treatment within 4 week prior to randomization with cyclosporine A or tacrolimus, everolimus, sirolimus (calcineurin or mammalian target of rapamycin (mTOR) inhibitors).
21. Treatment with cytochrome P3A (CYP3A) inducers within 4 weeks prior to randomization
22. Known hypersensitivity to drugs of the same class as the study drug, or any of their excipients.
23. Planned treatment, or treatment, with another investigational drug within 1 month prior to randomization.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2008-05; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loic Perchenet, PhD, Study Chair — Actelion
Locations (153):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialists, Pheonix, Arizona
  - GLVA Healthcare Center, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Liu Center for Pulmonary Hypertension, Torrance, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Emory University Hospital - McKelvey Center for Lung Transplantation & Pulmonary Vascular Disease, Atlanta, Georgia
  - Pulmonary & Critical Care of Atlanta, Atlanta, Georgia
  - Southeastern Lung Care, Decatur, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kentuckiana Pulmonary Associate, PLLC, Louisville, Kentucky
  - Medical Center of Louisiana at New Orleans, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Pulmonary/Critical Care Division/Tufts New England Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of NJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Columbia University Medical Center - Pediatric Cardiology, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Ohio Heart Health Center, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Medical Center - St. Paul University, Dallas, Texas
  - Baylor College of Medicine and the Methodist Hospital, Houston, Texas
  - Dept. of Pulmonary Medicine - Latter Day Saints Hospital, Salt Lake City, Utah
  - Sentara Hospital T/A Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Comprehensive Cardiovascular Care Group, Milwaukee, Wisconsin
- Argentina (8):
  - Fundacion Favaloro, Buenos Aires
  - Hospital Britanico, Buenos Aires
  - Sanatorio MITRE, Buenos Aires
  - SANATORIO OTAMENDI y MIROLI, Buenos Aires
  - Instituto Cardiologia Corrientes, Corrientes
  - Htal Italiano Cordoba, Córdoba
  - Htla privado de Cordoba, Córdoba
  - 'Hospital Italiano - Garibaldi de Rosario, Santa Fe
- Australia (3):
  - St. Vincent's Hospital, Darlinghurst, NSW
  - The Alfred Hospital, Melbourne, VIC
  - Royal Brisbane Hospital, Sunshine Coast
- Medical University of Vienna/ Department of Internal Medicine II, Division of Cardiology, Vienna, Austria
- Belarus (3):
  - Republican reserach - Pratical Centre of Cardilogy, Minsk
  - Minsk Regional Clinical Hospital, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- University Hospital Gasthuisberg / Kliniekhoofd, Interne Geneeskunde - I.G. Pneumologie, Leuven, Belgium
- Specialized Hospital for Active Treatment of Cardio-Vascular Diseases / Department of Pediatric Cardiology, Sofia, Bulgaria
- Canada (5):
  - London Health Sciences Centre / Victoria Hospital, London, Ontario
  - L'Hopital Laval, Saint-Foy, Quebec
  - Peter Lougheed Centre, Calgary
  - Toronto General Hospital, Toronto
  - Vancouver General Hospital, Vancouver
- Chile (3):
  - 'Pontificia Universidad Catolica de Chile, Santiago, Chile
  - Hospital del Torax, Santiago, Chile
  - Hospital San Juan de Dios, Santiago, Chile
- China (9):
  - Guangdong General Hospital, Cardiology Department, Guangzhou, Guangdong
  - Jiangsu Province Hospital - Pneumology Department, Nanjing, Jiangsu
  - Beijing Anzhen Hospital of the Capital University of Medical Sciences, Cardiology Department, Beijing
  - Peking Union Medcical College Hospital, Rheumatology Department, Beijing
  - Chinese PLA General Hospital (301 Hospital), Cardiology Department, Beijing
  - Renji Hospital, Rheumatology Dept, Shanghai
  - Zhongshan Hospital Fudan University, Cardiology Dept, Shanghai
  - Renji Hospital, Cardiology Dept, Shanghai
  - Shanghai Pulmonary Hospital, Dept of Pulmonary Circulation, Shanghai
- Colombia (2):
  - Fundación Clínica Shaio, Bogotá
  - 'Fundacion Cardiovascular de Colombia, Floridablanca, Santander
- Clinical Hospital Center, Rijeka, Croatia
- France (3):
  - Hôpital Antoine Béclère / Service de Pneumologie, Clamart
  - Hôpital Arnaud de Villeneuve Service des Maladies Respiratoires, Montpellier
  - Hopital Haut-Leveque - Maison du Haut-Leveque, Pessac
- Germany (12):
  - Unfallkrankenhaus Berlin, Klinik für Innere Medizin, Berlin
  - Universität zu Köln, Medizinische Klinik III, Abteilung Kardiologie, Cologne
  - Medizinische Klinik und Poliklinik I Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikums Gießen und Marburg GmbH / Medizinische Klinik und Poliklinik II, Innere Med., Giessen
  - Universität Greifswald / Klinik für Innere Medizin B,, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf / Onkologie, Hämatologie und Knochenmarktransplantation mit Sektion Pneumologie, Hamburg
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Universitätskliniken des Saarlandes / Medizinische Klinik und Poliklinik, Innere Medizin V, Homburg/Saar
  - Universtätsklinik Leipzig, Leipzig
  - Klinikum der Johannes Gutenberg-Universität / II. Medizinische Klinik und Poliklinik, Mainz
  - Medizinische Klinik und Poliklinik I der Ludwig-Maximilians-Universität München / Klinikum Großhadern, Schwerpunkt Pneumologie, Munich
  - Universitätsklinikum Regensburg / Innere Medizin II, Regensburg
- Hong Kong (2):
  - Prince of Wales Hospital/ Division of Rheumatology, Department of Medicine & Therapeutics, Hong Kong
  - Queen Mary Hospital / Division of Cardiology, Department of Medicine, Hong Kong
- Hungary (3):
  - Gottsegen György Országos Kardiológiai Intézet (Hungarian Institute of Cardiology), Budapest
  - Semmelweis University, Pulmonolgy Clinic, Budapest
  - University of Szeged Albert Szent-Györgyi Medical and Pharmaceutical Center, Faculty of General Medicine, II. Internal Medicine Clinic, Cardiology Center, Szeged
- India (6):
  - Life Care Institute of Medical Science & Research, Ahmedabad, Ahmedabad
  - G B Pant Hospital & Maulana Azad Medical College, Delhi
  - Care Hospital, Hyderabad
  - King Edward VII Memorial Hospital (KEM) Hospital, Mumbai
  - P D Hinduja National Hospital and Medical Research Centre/ Pulmunory Medicine, Mumbai
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
- Israel (5):
  - Lady Davis Carmel Medical Center / Department of Cardiovascular Medicine, Pulmonary Division, Haifa
  - Rabin Medical Center - Belinson campus - Pulmonary Institute, Petach - Tikvah
  - Pulmonary Institute, Kaplan Medical Center, Rehovot
  - Sourasky Medical Center - Division of Pulmonary Medicine and Allergy, Tel Aviv
  - The pulmonary institute Sheba Medical centre, Tel Litwinsky
- Policlinico Umberto I, Cardiologia, Roma, Italy
- Institut Jantung Negara (National Heart Institute), Kuala Lumpur, Malaysia
- Mexico (2):
  - 'Instituto Nacional de Cardiología (INC) Ignacio Chávez, Mexico City
  - Unidad de Investigación Clinica en Medicina, SC, Monterrey Nuevo León
- St. Antonius ziekenhuis, Nieuwegein, Netherlands
- Aker University Dept of Cardilogy, Oslo, Norway
- Peru (2):
  - Hospital Alberto Sabogal Sologuren - EsSALUD, Lima
  - IInstituto de Enfermedades Respiratorias, Clinica San Gabriel, Lima
- Poland (3):
  - Klinika Chorob Serca i Naczyn Instytut Kardiologii Collegium Medicum UJ, Krakow
  - Klinika Chorób Wewnętrznych Klatki Piersiowej, Warsaw
  - III Katedra i Oddział Kliniczny Kardiologii Slaskiego Uniwersytetu Medycznego, Zabrze
- Romania (2):
  - Institutul de boli cardiovasculare / Clinica de Cardiologie, Bucharest
  - Institutul de Pneumologie "Marius Nasta" / I. Clinica de Pneumoftiziologie, Bucharest
- Russia (10):
  - Municipal Health Care Institution "Kemerovo Cardiology Dispensary", Kemerovo
  - Federal State Institution "Scientific Research Institute of Pulmonology of Roszdrav", Moscow
  - State Health Care Institution of Moscow "City Clinical Hospital #1 named after N. I. Pirogov", Moscow
  - Federal State Institution "Russian Cardiology Scientific and Production Complex of Rosmedtechnology", Moscow
  - Federal State Institution "Federal Center of Heart, Blood and Endocrinology named after V.A. Almazov" of Rosmedtechnology, Saint Petersburg
  - State Educational Institution of High Professional Education, Saint Petersburg
  - State Institution "Scientific Research Institute of Cardiology" of Tomsk Scientific Center of RAMS, Siberian branch, Tomsk
  - Tomsk Regional Clinical Hospital / Pulmonology Unit, Tomsk
  - Municipal Health Care Institution "Clinical Hospital of Emergency Care named after N.V. Soloviov", Yaroslavl
  - Sverdlovsk Regional Clinical Hospital # 1/ Cardiology Department (2nd Therapy Department), Yekaterinburg
- Serbia (3):
  - University Children's Hospital (UNIVERZITETSKA DEČJA KLINIKA), Belgrade
  - University Clinical Center of Serbia / Institute for Lung Diseases and Tuberculosis, Belgrade
  - Zemun Clinical Hospital (Kliničko-bolnički centar "Zemun" ) / Department of Cardiology, Belgrade
- Singapore (2):
  - National University Hospital/ The Heart Institute, Singapore
  - Singapore General Hospital, Singapore
- Slovakia (2):
  - National Institute of Cardiovascular Diseases (Národný ústav srdcových a cievnych chorôb, a.s. - NÚSCH) / Department of Heart Transplantation, Bratislava
  - Slovak Medical University (Slovenská zdravotnícka univerzita) / Faculty of Medical Speciality Studies (Fakulta zdravotníckych špecializačných štúdií), Department of Cardiology and Angiology, Bratislava
- South Africa (4):
  - Netcare Milpark Hospital,Center for Chest Disease, Johannesburg
  - Chris Hani Baragwanath Hospital, Department of Cardiology, Johannesburg
  - Tread Research, Parow
  - Block 4, Vergelegen Medi-Clinic, Somerset West
- Spain (6):
  - Hospital Juan Canalejo Servicio de Neumología, A Coruña
  - Hospital Universitario Vall d'Hebron, Pneumology Unit, Planta Baja Hospital General, Barcelona
  - Hospital Clínico I Provincial, Servicio de Neumología., Barcelona
  - Hospital 12 Octubre/ Cardiology department Planta 5a., Madrid
  - Hospital Clínico Virgen de la Victoria / Pneumology Unit,, Málaga
  - Hospital Montecelo, Servicio de Neumología, Pontevedra
- Sweden (2):
  - University Hospital in Lund, Heart and Lung Division, Lund
  - Servicio de Medicina Interna, Unidad de Hipertensión Pulmonar, Uppsala
- Taiwan (2):
  - Taichung Veterans General Hospital / Division of Allergy, Immunology and Rheumatology, Taichung
  - National Taiwan University Hospital/ Thoracic Surgical Division, Surgical Department, Taipei
- Thailand (4):
  - Ramathibodi Hospital, Mahidol University, Cardiology Unit, Department of Medicine,, Bangkok
  - Siriraj Hospital/ Department of Pediatrics, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok
  - Chiang Mai Hospital / Division of Rheumatology, Department of Medicine, Faculty of Medicine, Chiang Mai University, Chiang Mai
  - Srinagarind Hospital/Division of Rheumatology, Department of Medicine, Faculty of Medicine, Khon Kaen University, Khon Kaen
- Istanbul University Cardiology Institure, Istanbul, Turkey (Türkiye)
- Ukraine (2):
  - Dnipropetrovsk State Medical Academy / Regional Diagnostic Center, Department of electrophysiologic researches and anaesthesiologic aid, Dnipro
  - Danylo Halytskyi Lviv State Medical University, Lviv
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Result] Pulido T, Adzerikho I, Channick RN, Delcroix M, Galie N, Ghofrani HA, Jansa P, Jing ZC, Le Brun FO, Mehta S, Mittelholzer CM, Perchenet L, Sastry BK, Sitbon O, Souza R, Torbicki A, Zeng X, Rubin LJ, Simonneau G; SERAPHIN Investigators. Macitentan and morbidity and mortality in pulmonary arterial hypertension. N Engl J Med. 2013 Aug 29;369(9):809-18. doi: 10.1056/NEJMoa1213917. PMID 23984728
- [Derived] Di Scala L, Bacchi M, Bayer B, Turricchia S. Adjusting Overall Survival Estimates of Macitentan in Pulmonary Arterial Hypertension After Treatment Switching: Results from the SERAPHIN Study. Adv Ther. 2022 Sep;39(9):4346-4358. doi: 10.1007/s12325-022-02253-8. Epub 2022 Aug 1. PMID 35917059
- [Derived] Souza R, Delcroix M, Galie N, Jansa P, Mehta S, Pulido T, Rubin L, Sastry BKS, Simonneau G, Sitbon O, Torbicki A, Boyanova N, Chamitava L, Stein C, Channick RN. Long-Term Safety, Tolerability and Survival in Patients with Pulmonary Arterial Hypertension Treated with Macitentan: Results from the SERAPHIN Open-Label Extension. Adv Ther. 2022 Sep;39(9):4374-4390. doi: 10.1007/s12325-022-02199-x. Epub 2022 Jul 12. PMID 35819570
- [Derived] Torbicki A, Bacchi M, Delcroix M, Farber HW, Ghofrani HA, Hennessy B, Jansa P, Mehta S, Perchenet L, Pulido T, Rosenberg D, Rubin LJ, Sastry BKS, Simonneau G, Sitbon O, Souza R, Wei LJ, Channick R, Benza R. Integrating Data From Randomized Controlled Trials and Observational Studies to Assess Survival in Rare Diseases. Circ Cardiovasc Qual Outcomes. 2019 May;12(5):e005095. doi: 10.1161/CIRCOUTCOMES.118.005095. PMID 31109190
- [Derived] Krause A, Zisowsky J, Dingemanse J. Modeling of pharmacokinetics, efficacy, and hemodynamic effects of macitentan in patients with pulmonary arterial hypertension. Pulm Pharmacol Ther. 2018 Apr;49:140-146. doi: 10.1016/j.pupt.2018.02.005. Epub 2018 Feb 28. PMID 29501590
- [Derived] McLaughlin VV, Hoeper MM, Channick RN, Chin KM, Delcroix M, Gaine S, Ghofrani HA, Jansa P, Lang IM, Mehta S, Pulido T, Sastry BKS, Simonneau G, Sitbon O, Souza R, Torbicki A, Tapson VF, Perchenet L, Preiss R, Verweij P, Rubin LJ, Galie N. Pulmonary Arterial Hypertension-Related Morbidity Is Prognostic for Mortality. J Am Coll Cardiol. 2018 Feb 20;71(7):752-763. doi: 10.1016/j.jacc.2017.12.010. PMID 29447737
- [Derived] Jansa P, Pulido T. Macitentan in Pulmonary Arterial Hypertension: A Focus on Combination Therapy in the SERAPHIN Trial. Am J Cardiovasc Drugs. 2018 Feb;18(1):1-11. doi: 10.1007/s40256-017-0260-1. PMID 29280064
- [Derived] Mehta S, Sastry BKS, Souza R, Torbicki A, Ghofrani HA, Channick RN, Delcroix M, Pulido T, Simonneau G, Wlodarczyk J, Rubin LJ, Jansa P, Hunsche E, Galie N, Perchenet L, Sitbon O. Macitentan Improves Health-Related Quality of Life for Patients With Pulmonary Arterial Hypertension: Results From the Randomized Controlled SERAPHIN Trial. Chest. 2017 Jan;151(1):106-118. doi: 10.1016/j.chest.2016.08.1473. Epub 2016 Sep 23. PMID 27671974
- [Derived] Simonneau G, Channick RN, Delcroix M, Galie N, Ghofrani HA, Jansa P, Le Brun FO, Mehta S, Perchenet L, Pulido T, Sastry BK, Sitbon O, Souza R, Torbicki A, Rubin LJ. Incident and prevalent cohorts with pulmonary arterial hypertension: insight from SERAPHIN. Eur Respir J. 2015 Dec;46(6):1711-20. doi: 10.1183/13993003.00364-2015. Epub 2015 Oct 22. PMID 26493786
- [Derived] Channick RN, Delcroix M, Ghofrani HA, Hunsche E, Jansa P, Le Brun FO, Mehta S, Pulido T, Rubin LJ, Sastry BKS, Simonneau G, Sitbon O, Souza R, Torbicki A, Galie N. Effect of macitentan on hospitalizations: results from the SERAPHIN trial. JACC Heart Fail. 2015 Jan;3(1):1-8. doi: 10.1016/j.jchf.2014.07.013. Epub 2014 Nov 11. PMID 25457902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 955 patients were screened from 158 centers in 39 countries, and 742 patients from 151 centers in 39 countries were randomized
Groups:
- Placebo: Matching ACT-064992 placebo tablet, once daily
- ACT-064992 3 mg: ACT-064992 tablet, 3 mg, once daily
- ACT-064992 10 mg: ACT-064992 tablet, 10 mg, once daily
Period: Overall Study
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg
Started | 250 | 250 | 242
Completed | 194 | 192 | 201
Not Completed | 56 | 58 | 41
Not completed — Death | 44 | 47 | 34
Not completed — Withdrawal of consent | 4 | 6 | 4
Not completed — Lost to Follow-up | 7 | 5 | 2
Not completed — Administrative reason | 0 | 0 | 1
Not completed — Incorrect randomization | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For the baseline measures of age, gender, and World Health Organization (WHO) functional class, data were missing for 1 patient in the placebo group and for 2 patients in the 3 mg macitentan group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg | Total
Number analyzed (Participants) | 250 | 250 | 242 | 742
Age, Categorical [Number; unit: participants]
  <=18 years | 7 | 7 | 6 | 20
  Between 18 and 65 years | 199 | 208 | 209 | 616
  >=65 years | 43 | 33 | 27 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (17.03) | 44.5 (16.26) | 45.5 (14.99) | 45.6 (16.13)
Gender [Number; unit: participants]
  Female | 184 | 187 | 194 | 565
  Male | 65 | 61 | 48 | 174
Region of Enrollment [Number; unit: participants]
  Argentina | 14 | 16 | 13 | 43
  Australia | 2 | 4 | 4 | 10
  Austria | 1 | 1 | 2 | 4
  Belarus | 7 | 8 | 8 | 23
  Belgium | 1 | 0 | 1 | 2
  Bulgaria | 1 | 3 | 2 | 6
  Canada | 7 | 5 | 4 | 16
  Chile | 9 | 10 | 9 | 28
  China | 31 | 29 | 27 | 87
  Colombia | 3 | 3 | 3 | 9
  Croatia | 0 | 0 | 1 | 1
  Denmark | 1 | 0 | 0 | 1
  France | 5 | 3 | 3 | 11
  Germany | 17 | 14 | 13 | 44
  Hong Kong | 1 | 2 | 1 | 4
  Hungary | 1 | 3 | 2 | 6
  India | 15 | 17 | 15 | 47
  Israel | 6 | 6 | 8 | 20
  Italy | 2 | 2 | 1 | 5
  Malaysia | 2 | 2 | 3 | 7
  Mexico | 13 | 13 | 14 | 40
  Netherlands | 0 | 1 | 0 | 1
  Norway | 1 | 0 | 1 | 2
  Peru | 3 | 2 | 2 | 7
  Poland | 7 | 7 | 7 | 21
  Romania | 5 | 5 | 6 | 16
  Russian Federation | 25 | 24 | 23 | 72
  Serbia | 7 | 5 | 4 | 16
  Singapore | 4 | 5 | 4 | 13
  Slovakia | 1 | 2 | 3 | 6
  South Africa | 9 | 7 | 8 | 24
  Spain | 4 | 5 | 6 | 15
  Sweden | 3 | 2 | 2 | 7
  Taiwan | 4 | 5 | 5 | 14
  Thailand | 9 | 7 | 9 | 25
  Turkey | 1 | 1 | 1 | 3
  United Kingdom | 1 | 1 | 3 | 5
  United States | 23 | 25 | 19 | 67
  Ukraine | 4 | 5 | 5 | 14
World Health Organisation Functional Class [Number; unit: participants] — Class I: no limitation of usual physical activity (PA) which does not increase dyspnea, fatigue, chest pain, or presyncope.
  Class II: mild limitation of PA. No discomfort at rest. Normal PA increases dyspnea, fatigue, chest pain, or presyncope.
  Class III: marked limitation of PA. No discomfort at rest. Less than ordinary activity increases dyspnea, fatigue, chest pain, or presyncope.
  Class IV: unable to perform any PA and who may have signs of right ventricular failure. Dyspnea and/or fatigue may be present at rest and symptoms are increased by almost any PA.
  participants
    Class I | 0 | 0 | 1 | 1
    Class II | 129 | 138 | 120 | 387
    Class III | 116 | 105 | 116 | 337
    Class IV | 4 | 5 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Time to First Confirmed Morbidity or Mortality Event up to the End of Treatment (Kaplan-Meier Estimate of Patients Without a Morbidity or Mortality Event)
Description: Morbidity or mortality events were defined as: a) Death; b) Atrial septostomy; c) Lung transplantation; d) Initiation of intravenous (i.v.) or subcutaneous prostanoids, or; e) Other worsening of pulmonary arterial hypertension (PAH).
  Other worsening of PAH was defined by the combined occurrence of all the following 3 events:
  At least 15% decrease in the 6 minute walk distance from baseline, confirmed by 2 tests performed on separate days, within 2 weeks.
  AND worsening of PAH symptoms including at least one of the following:
  a) Increase in WHO Functional Class (WHO FC), or no change in patients in WHO FC IV at baseline; b) Appearance or worsening of signs of right heart failure that did not respond to optimized oral diuretic therapy
  AND need for new treatment(s) for PAH that included the following: a) Oral or inhaled prostanoids; b) Oral phosphodiesterase inhibitors; c) Endothelin receptor antagonists (only after discontinuation of study treatment; d) i.v. diuretics
Time Frame: Up to end of treatment (data presented up to month 36)
Population: All randomized patients
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg
Number analyzed (Participants) | 250 | 250 | 242
percentage of participants-Kaplan Meier
  Kaplan-Meier estimate at Month 6 | 80.1 | 89.3 | 92.7
  Kaplan-Meier estimate at Month 12 | 71.4 | 81.6 | 85.5
  Kaplan-Meier estimate at Month 18 | 61.5 | 72.5 | 79.9
  Kaplan-Meier estimate at Month 24 | 57.3 | 65.5 | 74.3
  Kaplan-Meier estimate at Month 30 | 50.2 | 61.9 | 70.0
  Kaplan-Meier estimate at Month 36 | 47.0 | 55.0 | 63.2
Statistical Analysis 1: Comparison: Placebo vs ACT-064992 3 mg; Test type: Superiority or Other; p = 0.0108, Log Rank; Hazard Ratio (HR) = 0.704, 97.5% CI 2-sided [0.516 to 0.960]
Statistical Analysis 2: Comparison: Placebo vs ACT-064992 10 mg; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.547, 97.5% CI 2-sided [0.392 to 0.762]

2. Secondary Outcome: Time to Death Due to PAH or Hospitalisation for PAH up to the End of Treatment (Kaplan-Meier Estimate of Patients Without an Event)
Description: Events of PAH or hospitalization for PAH up to the end of treatment included: death due to PAH, or onset of a treatment-emergent adverse event with a fatal outcome due to PAH occurring up to 4 weeks after the end of treatment, or hospitalisation for PAH up to the end of treatment.
Time Frame: Up to end of treatment (data presented up to month 36)
Population: All randomized patients
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg
Number analyzed (Participants) | 250 | 250 | 242
percentage of participants-Kaplan Meier
  Kaplan-Meier Estimate at Month 6 | 84.8 | 90.8 | 94.6
  Kaplan-Meier Estimate at Month 12 | 76.7 | 84.9 | 89.8
  Kaplan-Meier Estimate at Month 18 | 69.0 | 78.1 | 84.8
  Kaplan-Meier Estimate at Month 24 | 67.9 | 75.1 | 81.7
  Kaplan-Meier Estimate at Month 30 | 62.0 | 70.3 | 77.9
  Kaplan-Meier Estimate at Month 36 | 55.4 | 67.1 | 70.6
Statistical Analysis 1: Comparison: Placebo vs ACT-064992 3 mg; Test type: Superiority or Other; p = 0.0146, Log Rank; Hazard Ratio (HR) = 0.669, 97.5% CI 2-sided [0.462 to 0.970]
Statistical Analysis 2: Comparison: Placebo vs ACT-064992 10 mg; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.500, 97.5% CI 2-sided [0.335 to 0.747]

3. Secondary Outcome: Time to Death Due to Any Cause up to the End of Treatment (Kaplan-Meier Estimate of Patients Without an Event)
Description: Events of death due to any cause up to the end of treatment (plus 7 days)
Time Frame: Up to end of treatment (data presented up to month 36)
Population: All randomized patients
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg
Number analyzed (Participants) | 250 | 250 | 242
percentage of participants-Kaplan Meier
  Kaplan-Meier Estimate at Month 6 | 95.2 | 97.1 | 97.4
  Kaplan-Meier Estimate at Month 12 | 93.6 | 95.6 | 96.4
  Kaplan-Meier Estimate at Month 18 | 92.4 | 94.6 | 94.8
  Kaplan-Meier Estimate at Month 24 | 91.7 | 91.7 | 94.8
  Kaplan-Meier Estimate at Month 30 | 89.8 | 89.9 | 93.3
  Kaplan-Meier Estimate at Month 36 | 89.8 | 87.3 | 93.3
Statistical Analysis 1: Comparison: Placebo vs ACT-064992 3 mg; Test type: Superiority or Other; p = 0.9249, Log Rank; Hazard Ratio (HR) = 0.971, 97.5% CI 2-sided [0.477 to 1.976]
Statistical Analysis 2: Comparison: Placebo vs ACT-064992 10 mg; Test type: Superiority or Other; p = 0.2037, Log Rank; Hazard Ratio (HR) = 0.638, 97.5% CI 2-sided [0.287 to 1.418]

4. Secondary Outcome: Time to Death Due to Any Cause up to the End of Study (Kaplan-Meier Estimate of Patients Without an Event)
Description: Events of death due to any cause up to the end of study (EOS). The initiation of EOS procedure occurred when the target of 285 events was expected to have been achieved (30 January 2012).
Time Frame: Up to end of study (data presented up to month 36)
Population: All randomized patients
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg
Number analyzed (Participants) | 250 | 250 | 242
percentage of participants-Kaplan Meier
  Kaplan-Meier Estimate at Month 6 | 94.7 | 96.4 | 96.3
  Kaplan-Meier Estimate at Month 12 | 91.4 | 93.9 | 95.0
  Kaplan-Meier Estimate at Month 18 | 89.3 | 91.4 | 93.3
  Kaplan-Meier Estimate at Month 24 | 87.2 | 87.3 | 89.1
  Kaplan-Meier Estimate at Month 30 | 82.6 | 83.4 | 86.9
  Kaplan-Meier Estimate at Month 36 | 80.7 | 80.0 | 82.9
Statistical Analysis 1: Comparison: Placebo vs ACT-064992 3 mg; Test type: Superiority or Other; p = 0.8312, Log Rank; Hazard Ratio (HR) = 1.046, 97.5% CI 2-sided [0.653 to 1.673]
Statistical Analysis 2: Comparison: Placebo vs ACT-064992 10 mg; Test type: Superiority or Other; p = 0.2509, Log Rank; Hazard Ratio (HR) = 0.771, 97.5% CI 2-sided [0.464 to 1.282]

5. Secondary Outcome: Change From Baseline to Month 6 in 6-minute Walk Distance
Description: The 6-minute walk test (6MWT) is a non-encouraged test, performed in a 30 m long flat corridor, where the patient is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. These guidelines were provided to all sites. For patients who had never performed a 6MWT previously, a training test was required before the qualifying tests for inclusion were performed.
Time Frame: Baseline to month 6
Population: All randomized patients excluding 1 patient in the placebo group who did not start study treatment and 2 patients in the ACT-064992 3 mg group who did not follow appropriate consent procedures and were not included in the analysis
Measure: Mean (Standard Deviation); unit: metres
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg
Number analyzed (Participants) | 249 | 248 | 242
metres
  Baseline | 352 (110.6) | 364 (95.5) | 363 (93.2)
  Change from baseline at Month 6 | -9.4 (100.59) | 7.4 (93.15) | 12.5 (83.54)

6. Secondary Outcome: Number of Patients With Improvements in World Health Organization Functional Class From Baseline to Month 6
Description: Class I: no limitation of usual physical activity (PA) which does not increase dyspnea, fatigue, chest pain, or presyncope.
  Class II: mild limitation of PA. No discomfort at rest. Normal PA increases dyspnea, fatigue, chest pain, or presyncope.
  Class III: marked limitation of PA. No discomfort at rest. Less than ordinary activity increases dyspnea, fatigue, chest pain, or presyncope.
  Class IV: unable to perform any PA and who may have signs of right ventricular failure. Dyspnea and/or fatigue may be present at rest and symptoms are increased by almost any PA.
Time Frame: Baseline to month 6
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg
Number analyzed (Participants) | 249 | 248 | 242
participants | 32 | 49 | 54

7. Secondary Outcome: Pulmonary Vascular Resistance at Baseline and Month 6
Description: In a sub-study, hemodynamic variables were assessed at baseline and Month 6. If the patient had undergone a right heart catheterization during the 3 months prior to randomization, these results were to be used as baseline values, if the background therapy had not changed during the intervening period.
Time Frame: Baseline to month 6
Population: All randomized patients participating in the pharmacokinetic/pharmacodynamic sub-study
Measure: Mean (Full Range); unit: (dyn*sec/cm^5)
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg
Number analyzed (Participants) | 50 | 47 | 48
(dyn*sec/cm^5)
  Baseline | 886 (587) [259 to 3390] | 945 (541) [250 to 2317] | 907 (550) [254 to 2279]
  Month 6 | 1042 (656) [164 to 3409] | 736 (434) [71 to 2308] | 680 (497) [158 to 2813]

8. Secondary Outcome: Cardiac Index at Baseline and Month 6
Description: as for outcome 7
Time Frame: Baseline to month 6
Population: All randomized patients participating in the pharmacokinetic/pharmacodynamic sub-study
Measure: Mean (Full Range); unit: L/min/m^2
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg
Number analyzed (Participants) | 50 | 47 | 48
L/min/m^2
  Baseline | 2.54 [1.31 to 4.54] | 2.34 [1.13 to 5.15] | 2.63 [1.20 to 6.24]
  Month 6 | 2.21 [1.06 to 3.89] | 2.69 [1.26 to 5.59] | 2.93 [1.46 to 5.11]
  Change from Baseline to Month 6 | -0.33 [-2.53 to 0.44] | 0.36 [-0.81 to 1.76] | 0.30 [-2.97 to 1.99]

9. Other Pre Specified Outcome: Summary of the First Causes of Morbidity or Mortality
Description: as for outcome 1
Time Frame: Up to end of treatment (Up to 36 months)
Population: All randomized patients
Measure: Number; unit: participants
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg
Number analyzed (Participants) | 250 | 250 | 242
participants
  Other worsening of PAH | 93 | 72 | 59
  Death | 17 | 21 | 16
  Prostanoid initiation (i.v. or s.c.) | 6 | 1 | 1
  Lung transplantation | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to end of treatment plus 28 days (Up to approximately 36 months)
Description: One patient in the placebo group never received study treatment and was not included in the analysis. Adverse events during treatment period and up to 28 days after treatment discontinuation
Arm/Group | Placebo | ACT-064992 3 mg | ACT-064992 10 mg
Serious Adverse Events (participants affected / at risk) | 137/249 | 130/250 | 109/242
Other Adverse Events (participants affected / at risk) | 219/249 | 227/250 | 222/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=249) | ACT-064992 3 mg (N=250) | ACT-064992 10 mg (N=242)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 56 | 48 | 32
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 3
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PHARYNGEAL CYST (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 40 | 21 | 23
ATRIAL FLUTTER (Cardiac disorders) | 2 | 2 | 4
CARDIAC ARREST (Cardiac disorders) | 1 | 3 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1 | 2
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1 | 1
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 | 1 | 1
BRADYCARDIA (Cardiac disorders) | 0 | 1 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 1 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 3 | 0 | 1
ACUTE RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 1 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 1 | 0
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 1 | 0
PALPITATIONS (Cardiac disorders) | 0 | 1 | 0
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0 | 0
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 | 0 | 0
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0
TACHYARRHYTHMIA (Cardiac disorders) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 8 | 7 | 4
GASTROENTERITIS (Infections and infestations) | 2 | 3 | 2
BRONCHITIS (Infections and infestations) | 1 | 2 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 3 | 0
URINARY TRACT INFECTION (Infections and infestations) | 3 | 0 | 2
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 2 | 0
ERYSIPELAS (Infections and infestations) | 0 | 2 | 0
SEPSIS (Infections and infestations) | 4 | 0 | 1
LUNG INFECTION (Infections and infestations) | 1 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 1 | 0
WOUND INFECTION (Infections and infestations) | 1 | 0 | 1
BACTERIAL SEPSIS (Infections and infestations) | 0 | 0 | 1
BRONCHITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1
DENGUE FEVER (Infections and infestations) | 0 | 1 | 0
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 | 1 | 0
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 | 1 | 0
HEPATITIS E (Infections and infestations) | 0 | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1 | 0
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 0
OMPHALITIS (Infections and infestations) | 0 | 0 | 1
OVERGROWTH BACTERIAL (Infections and infestations) | 0 | 0 | 1
PAROTID ABSCESS (Infections and infestations) | 0 | 0 | 1
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 | 1 | 0
PNEUMONIA MORAXELLA (Infections and infestations) | 0 | 1 | 0
PNEUMONIA NECROTISING (Infections and infestations) | 0 | 0 | 1
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 | 1 | 0
POST PROCEDURAL CELLULITIS (Infections and infestations) | 0 | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 1
SALPINGO-OOPHORITIS (Infections and infestations) | 0 | 0 | 1
SIALOADENITIS (Infections and infestations) | 0 | 0 | 1
TRACHEOBRONCHITIS (Infections and infestations) | 0 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 1 | 0
VULVAL ABSCESS (Infections and infestations) | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 2 | 0 | 0
ABSCESS INTESTINAL (Infections and infestations) | 1 | 0 | 0
APPENDICITIS (Infections and infestations) | 1 | 0 | 0
CUTANEOUS TUBERCULOSIS (Infections and infestations) | 1 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0 | 0
INFECTED SKIN ULCER (Infections and infestations) | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 1 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 3 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 2
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1 | 1
ASCITES (Gastrointestinal disorders) | 1 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1
ANAL POLYP (Gastrointestinal disorders) | 0 | 0 | 1
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 0 | 0 | 1
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0
MALABSORPTION (Gastrointestinal disorders) | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 0
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
PANCREATITIS RELAPSING (Gastrointestinal disorders) | 0 | 0 | 1
PEPTIC ULCER (Gastrointestinal disorders) | 0 | 0 | 1
TONGUE HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 1 | 0
ILEUS (Gastrointestinal disorders) | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0
PANCREATIC MASS (Gastrointestinal disorders) | 1 | 0 | 0
PERITONITIS (Gastrointestinal disorders) | 1 | 0 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 1 | 4 | 3
SUDDEN DEATH (General disorders) | 0 | 1 | 2
SUDDEN CARDIAC DEATH (General disorders) | 2 | 1 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 1 | 1
PYREXIA (General disorders) | 0 | 2 | 0
ADVERSE DRUG REACTION (General disorders) | 1 | 1 | 0
DEATH (General disorders) | 1 | 0 | 1
CHEST DISCOMFORT (General disorders) | 0 | 1 | 0
DEVICE MALFUNCTION (General disorders) | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 1
MULTI-ORGAN DISORDER (General disorders) | 0 | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 0 | 1
DEVICE DISLOCATION (General disorders) | 1 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 6 | 7 | 4
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 0 | 1
SCIATICA (Nervous system disorders) | 0 | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 1 | 0
PRESYNCOPE (Nervous system disorders) | 2 | 0 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 0
TRIGEMINAL NEURALGIA (Nervous system disorders) | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 5 | 6
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 1
COAGULOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1
HYPOCOAGULABLE STATE (Blood and lymphatic system disorders) | 0 | 1 | 0
ANAEMIA MEGALOBLASTIC (Blood and lymphatic system disorders) | 1 | 0 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
OVARIAN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
ANGIOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
RECTOSIGMOID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
TONGUE NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 2 | 1
DYSFUNCTIONAL UTERINE BLEEDING (Reproductive system and breast disorders) | 0 | 2 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 1 | 1
METRORRHAGIA (Reproductive system and breast disorders) | 0 | 1 | 0
PELVIC FLUID COLLECTION (Reproductive system and breast disorders) | 0 | 0 | 1
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 1
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 2
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 | 0 | 2
HEPATIC ENZYME INCREASED (Investigations) | 0 | 1 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1 | 0
HEPATITIS B VIRUS TEST POSITIVE (Investigations) | 0 | 0 | 1
HIV TEST POSITIVE (Investigations) | 0 | 0 | 1
INTERNATIONAL NORMALISED RATIO DECREASED (Investigations) | 0 | 1 | 0
TRANSAMINASES INCREASED (Investigations) | 0 | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 | 1 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 1 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 0
BRAIN HERNIATION (Injury, poisoning and procedural complications) | 1 | 0 | 0
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0 | 0
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
TRAUMATIC BRAIN INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
SYSTEMIC SCLEROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 4 | 1
GLOMERULONEPHRITIS (Renal and urinary disorders) | 0 | 0 | 1
LUPUS NEPHRITIS (Renal and urinary disorders) | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1 | 0
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 | 1 | 0
CALCULUS URINARY (Renal and urinary disorders) | 1 | 0 | 0
PROTEINURIA (Renal and urinary disorders) | 1 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 1
HEPATITIS (Hepatobiliary disorders) | 1 | 0 | 1
JAUNDICE (Hepatobiliary disorders) | 1 | 1 | 0
BILIARY COLIC (Hepatobiliary disorders) | 0 | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 0 | 1 | 0
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 0 | 1 | 0
LIVER INJURY (Hepatobiliary disorders) | 0 | 1 | 0
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 | 0 | 0
POST CHOLECYSTECTOMY SYNDROME (Hepatobiliary disorders) | 1 | 0 | 0
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 2 | 5 | 0
COMPLICATION OF PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
HYPOTENSION (Vascular disorders) | 3 | 1 | 1
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 | 1 | 0
ARTERIOVENOUS FISTULA (Vascular disorders) | 0 | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 0 | 1
ARTERIAL THROMBOSIS (Vascular disorders) | 1 | 0 | 0
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 0 | 0
VASCULITIS NECROTISING (Vascular disorders) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 0 | 1
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0 | 0
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0 | 0
GOUT (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 1 | 0
ALCOHOLISM (Psychiatric disorders) | 0 | 1 | 0
MENTAL DISORDER (Psychiatric disorders) | 0 | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1 | 0
DRUG ABUSE (Psychiatric disorders) | 1 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
LEUKOCYTOCLASTIC VASCULITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PURPURA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 | 0 | 1
CARDIAC PACEMAKER INSERTION (Surgical and medical procedures) | 0 | 1 | 0
HEART AND LUNG TRANSPLANT (Surgical and medical procedures) | 0 | 1 | 0
TOOTH EXTRACTION (Surgical and medical procedures) | 1 | 0 | 0
GLYCOGEN STORAGE DISEASE TYPE V (Congenital, familial and genetic disorders) | 0 | 1 | 0
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 | 0 | 1
GLAUCOMA (Eye disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=249) | ACT-064992 3 mg (N=250) | ACT-064992 10 mg (N=242)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 32 | 48 | 37
OEDEMA PERIPHERAL (General disorders) | 45 | 40 | 44
NASOPHARYNGITIS (Infections and infestations) | 26 | 37 | 34
HEADACHE (Nervous system disorders) | 22 | 33 | 32
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 33 | 29 | 27
DIZZINESS (Nervous system disorders) | 27 | 24 | 26
ANAEMIA (Blood and lymphatic system disorders) | 7 | 18 | 30
BRONCHITIS (Infections and infestations) | 13 | 19 | 27
COUGH (Respiratory, thoracic and mediastinal disorders) | 30 | 20 | 21
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 21 | 24 | 16
CHEST PAIN (General disorders) | 19 | 18 | 17
DIARRHOEA (Gastrointestinal disorders) | 16 | 14 | 21
URINARY TRACT INFECTION (Infections and infestations) | 11 | 16 | 19
INSOMNIA (Psychiatric disorders) | 10 | 17 | 17
HYPOKALAEMIA (Metabolism and nutrition disorders) | 14 | 13 | 14
HYPOTENSION (Vascular disorders) | 8 | 13 | 14
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 18 | 16 | 10
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9 | 15 | 11
PHARYNGITIS (Infections and infestations) | 7 | 11 | 15
PALPITATIONS (Cardiac disorders) | 13 | 13 | 12
INFLUENZA (Infections and infestations) | 4 | 11 | 14
BACK PAIN (Musculoskeletal and connective tissue disorders) | 21 | 15 | 9
NAUSEA (Gastrointestinal disorders) | 13 | 12 | 12
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 9 | 9 | 15
SYNCOPE (Nervous system disorders) | 17 | 15 | 8
FATIGUE (General disorders) | 15 | 11 | 8
VOMITING (Gastrointestinal disorders) | 17 | 7 | 10
DYSPEPSIA (Gastrointestinal disorders) | 14 | 10 | 7
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 14 | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less